CLINICAL TRIAL: NCT00390884
Title: Safety and Immunogenicity of Fluzone® Influenza Virus Vaccine (2006-2007 Formulation) Among Healthy Children Immunized in Fall 2005 With Fluzone Vaccine or Placebo
Brief Title: Safety and Immunogenicity of Fluzone® Vaccine in Children Who Received 2 Doses of the 2005-2006 Fluzone Formulation.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: GRC29
Record Dates: First submitted 2006-10-20; First posted 2006-10-23 (Estimated); Results first posted 2009-12-31 (Estimated); Last update posted 2016-04-14 (Estimated); Status verified 2016-04

CONDITIONS: Influenza
Keywords: Fluzone®; Influenza; Influenza virus infection; Influenza vaccine
MeSH Terms: conditions — Influenza, Human | interventions — Influenza Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fluzone®-Primed Group (Experimental): Participants had received two doses of the 2005-2006 formulation of Fluzone® vaccine in the fall of 2005 (Study GRC28, NCT00242424), will receive 2 doses of Fluzone® Pediatric 2006-2007 formulation.
  Interventions: Biological: Influenza Virus Vaccine, Fluzone®
- Fluzone®-Naive Group (Experimental): Participants had never received Influenza vaccine and had received two doses of placebo in the fall of 2005 (Study GRC28, NCT00242424), will receive 2 doses of Fluzone® Pediatric 2006-2007 formulation.
  Interventions: Biological: Influenza Virus Vaccine, Fluzone®

INTERVENTIONS:
Biological: Influenza Virus Vaccine, Fluzone® — 0.25 mL, Intramuscular
  Other Names: Fluzone®
  Arms: Fluzone®-Primed Group
Biological: Influenza Virus Vaccine, Fluzone® — 0.25 mL, Intramuscular
  Other Names: Fluzone®
  Arms: Fluzone®-Naive Group

SUMMARY:
To compare the groups with respect to influenza immune responses following Dose 1 of Fluzone vaccine (2006-2007 formulation).

ELIGIBILITY:
Inclusion Criteria :

* Previously enrolled in study GRC28 and received 2 vaccinations of the assigned lot.
* Considered to be in good health on the basis of reported medical history and history-directed physical evaluation.
* Available for the duration of the study.
* Parent/legal representative willing and able to provide informed consent.
* Parent/legal representative able to attend all scheduled visits and comply with all trial procedures.
* Parent/legal representative willing to permit venipuncture for purposes of collecting a blood sample.

Exclusion Criteria :

* Receipt of any vaccine within the past 7 days (subjects may be deferred until after the seven days has passed.)
* Reported allergy to egg proteins, chicken proteins or any other constituent of the vaccine.
* Ever received any influenza vaccine, other than at Visits 1 and 2 of study GRC28, or known to have ever been diagnosed with laboratory-confirmed influenza.
* An acute illness with fever (rectal temperature ≥ 100.4°F [38.0°C]) in the 72 hours preceding enrollment in the trial (defer enrollment).
* Known bleeding disorder.
* Participation in any other interventional clinical trial within 30 days prior to enrollment, or planned participation in another interventional clinical trial prior to termination of the subject's participation in the study.
* Known or suspected impairment of immunologic function or receipt of immunosuppressive therapy or immunoglobulin since birth.
* Personal or immediate family history of congenital immune deficiency.
* Developmental delay, neurologic disorder, or seizure disorder.
* Chronic medical, congenital, or developmental disorder that, in the opinion of the investigator, could interfere with trial conduct or completion.
* Known Human Immunodeficiency Virus (HIV)-positive mother or Hepatitis B surface antigen (HBsAg)-positive mother.
* Known HIV, Hepatitis B, or Hepatitis C infection.
* Administration of immune globulin or other blood products within the last three months, or injected or oral corticosteroids or other immunomodulator therapy within six weeks of the study vaccine. Individuals on a tapering dose schedule of oral steroids lasting < 7 days may be included in the trial as long as they have not received more than one course within the last two weeks prior to enrollment.
* Prior personal history of Guillain-Barré syndrome.
* Any condition that, in the opinion of the investigator, would pose a health risk to the subject or interfere with the evaluation of the vaccine.

Ages: 11 Months to 14 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 173 (Actual)
Dates: Start 2006-10; Primary Completion 2007-06 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — sanofi pasteur Inc
Locations (5):
- United States (5):
  - Layton, Utah
  - Pleasant Grove, Utah
  - Provo, Utah
  - Salt Lake City, Utah
  - South Jordan, Utah

REFERENCES:
- See also: Related Info — http://www.sanofipasteur.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled into this study from 03 October 2006 to 04 January 2007 at 5 US clinical centers.
Pre-assignment Details: A total of 173 participants were enrolled, vaccinated, and analyzed.
Groups:
- Fluzone®-Primed Group: Participants had received two doses of the 2005-2006 formulation of Fluzone® vaccine in the fall of 2005 (Study GRC28 NCT00242424); they received two doses of Fluzone® Pediatric 2006-2007 formulation.
- Fluzone®-Naive Group: Participants had never received influenza vaccine and had received two doses of placebo (Study GRC28 NCT00242424); they received two doses of Fluzone® Pediatric 2006-2007 formulation.
Period: Overall Study
Arm/Group | Fluzone®-Primed Group | Fluzone®-Naive Group
Started | 116 | 57
Completed | 114 | 55
Not Completed | 2 | 2
Not completed — Withdrawal by Subject | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Fluzone®-Primed Group | Fluzone®-Naive Group | Total
Number analyzed (Participants) | 116 | 57 | 173
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 116 | 57 | 173
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: Months] | 13.8 (1.01) | 13.9 (1.13) | 13.8 (1.07)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48 | 22 | 70
  Male | 68 | 35 | 103
Region of Enrollment [Number; unit: participants]
  United States | 116 | 57 | 173

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Seroprotected Participants Post-vaccination With Fluzone®
Description: Seroprotection was defined as a Post-vaccination Hemagglutination Inhibition titer of greater than or equal to 1:40.
Time Frame: Day 28 Post-vaccination
Population: Hemagglutination inhibition titers to the Fluzone® vaccine antigens were assessed in the per-protocol immunogenicity population.
Measure: Number; unit: Percentage of Participants
Arm/Group | Fluzone®-Primed Group | Fluzone®-Naive Group
Number analyzed (Participants) | 94 | 50
Percentage of Participants
  Flu A/New Caledonia/20/99 (H1N1) Post-Dose 1 | 59 | 34
  Flu A/Wisconsin/67/2005 (H3N2) Post -Dose 1 | 95 | 80
  Flu B/Malaysia/2506/2004 Post-Dose 1 | 10 | 6
  Flu A/New Caledonia/20/99 (H1N1) Post-Dose 2 | 62 | 82
  Flu A/Wisconsin/67/2005 (H3N2) Post -Dose 2 | 79 | 94
  Flu B/Malaysia/2506/2004 Post-Dose 2 | 50 | 65

2. Secondary Outcome: Geometric Mean Titers (GMTs) of Hemagglutination Inhibition Antibodies Post-vaccination With Fluzone®
Description: Antibodies against Influenza virus in Fluzone® Vaccine determined by the Hemagglutination inhibition (HAI) assay method.
Time Frame: Day 28 Post-vaccination
Population: The Geometric Mean Titers were analyzed in the per-protocol immunogenicity population
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Fluzone®-Primed Group | Fluzone®-Naive Group
Number analyzed (Participants) | 94 | 50
Titers
  Flu A/New Caledonia/20/99 (H1N1) Post-Dose 1 | 41.3 [32.9 to 52.0] | 22.7 [17.9 to 28.7]
  Flu A/Wisconsin/67/2005 (H3N2) Post-Dose 1 | 144 [116 to 179] | 89.4 [55.4 to 144]
  Flu B/Malaysia/2506/2004 Post-Dose 1 | 11.1 [8.45 to 14.6] | 9.27 [6.31 to 13.6]
  Flu A/New Caledonia/20/99 (H1N1) Post-Dose 2 | 42.1 [27.3 to 64.8] | 78.4 [47.1 to 131]
  Flu A/Wisconsin/67/2005 (H3N2) Post-Dose 2 | 103 [68.9 to 155] | 217 [122 to 388]
  Flu B/Malaysia/2506/2004 Post-Dose 2 | 39.2 [25.5 to 60.3] | 63.9 [34.9 to 117]

3. Other Pre Specified Outcome: Percentage of Participants With At Least One Solicited Injection Site or Systemic Reaction Post-vaccination With Fluzone®
Description: Solicited injection site: tenderness, erythema, and swelling; Solicited systemic reactions: fever, vomiting, abnormal crying, drowsiness, appetite loss, and irritability, after each vaccination
Time Frame: Days 0-7 Post-vaccination
Population: The safety analysis was on all enrolled and vaccinated participants, intent-to-treat population.
Measure: Number; unit: Percentage of Participants
Arm/Group | Fluzone®-Primed Group | Fluzone®-Naive Group
Number analyzed (Participants) | 116 | 57
Percentage of Participants
  Any Injection Site Reaction Post-Dose 1 | 51 | 55
  Any Tenderness | 46 | 55
  Grade 3 Tenderness (Crying when limb is moved) | 0 | 0
  Any Redness (> 0.5 cm) | 7 | 7
  Grade 3 Redness (≥ 5.0 cm) | 0 | 0
  Any Swelling (> 0.5 cm) | 5 | 7
  Grade 3 Swelling (≥ 5.0 cm) | 0 | 0
  Any Injection Site Reaction Post-Dose 2 | 57 | 51
  Any Tenderness | 56 | 49
  Grade 3 Tenderness (Crying when limb is moved) | 1 | 0
  Any Redness (> 0.5 cm) | 7 | 6
  Grade 3 Redness (≥ 5.0 cm) | 0 | 0
  Any Swelling (> 0.5 cm) | 4 | 0
  Grade 3 Swelling (≥ 5.0 cm) | 0 | 0
  Any Injection Site Reaction - Any Dose | 68 | 69
  Any Tenderness | 65 | 69
  Grade 3 Tenderness (Crying when limb is moved) | 1 | 0
  Any Redness (> 0.5 cm) | 13 | 11
  Grade 3 Redness (≥ 5.0 cm) | 0 | 0
  Any Swelling (> 0.5 cm) | 6 | 7
  Grade 3 Swelling (≥ 5.0 cm) | 0 | 0
  Any Systemic Reaction Post-Dose 1 | 75 | 76
  Any Fever | 16 | 11
  Grade 3 Fever (≥ 103.2 ºF) | 0 | 0
  Any Vomiting | 13 | 16
  Grade 3 Vomiting (≥ 6 episodes per 24 hours) | 0 | 0
  Any Abnormal Crying | 42 | 36
  Grade 3 Abnormal Crying (> 3 hours) | 0 | 0
  Any Drowsiness | 32 | 31
  Grade 3 Drowsiness (Slept most of time) | 0 | 2
  Any Loss of Appetite | 38 | 33
  Grade 3 Loss of Appetite (Refuses ≥ 3 feeds) | 2 | 2
  Any Irritability | 66 | 64
  Grade 3 Irritability (Inconsolable) | 2 | 0
  Any Systemic Reaction Post-Dose 2 | 72 | 71
  Any Fever | 17 | 15
  Grade 3 Fever (≥ 103.2 ºF) | 2 | 2
  Any Vomiting | 12 | 16
  Grade 3 Vomiting (≥ 6 episodes per 24 hours) | 2 | 0
  Any Abnormal Crying | 39 | 33
  Grade 3 Abnormal Crying (> 3 hours) | 3 | 0
  Any Drowsiness | 32 | 33
  Grade 3 Drowsiness (Slept most of time) | 1 | 0
  Any Loss of Appetite | 32 | 33
  Grade 3 Loss of Appetite (Refuses ≥ 3 feeds) | 5 | 0
  Any Irritability | 57 | 60
  Grade 3 Irritability (Inconsolable) | 4 | 0
  Any Systemic Reaction - Any Dose | 88 | 89
  Any Fever | 29 | 24
  Grade 3 Fever (≥ 103.2 ºF) | 2 | 2
  Any Vomiting | 21 | 29
  Grade 3 Vomiting (≥ 6 episodes per 24 hours) | 2 | 0
  Any Abnormal Crying | 55 | 53
  Grade 3 Abnormal Crying (> 3 hours) | 3 | 0
  Any Drowsiness | 46 | 47
  Grade 3 Drowsiness (Slept most of time) | 1 | 2
  Any Loss of Appetite | 53 | 51
  Grade 3 Loss of Appetite (Refuses ≥ 3 feeds) | 5 | 2
  Any Irritability | 74 | 78
  Grade 3 Irritability (Inconsolable) | 5 | 0

ADVERSE EVENTS:
Time Frame: Adverse event data were collected for 2 months post-vaccination.
Arm/Group | Fluzone®-Primed Group | Fluzone®-Naive Group
Serious Adverse Events (participants affected / at risk) | 1/116 | 0/57
Other Adverse Events (participants affected / at risk) | 87/116 | 40/57
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fluzone®-Primed Group (N=116) | Fluzone®-Naive Group (N=57)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fluzone®-Primed Group (N=116) | Fluzone®-Naive Group (N=57)
Diarrhoea (Gastrointestinal disorders) | 23 (27) | 13 (14)
Teething (Gastrointestinal disorders) | 20 (30) | 5 (6)
Vomiting (Gastrointestinal disorders) | 17 (17) | 5 (5)
Pyrexia (General disorders) | 19 (20) | 11 (12)
Croup infectious (Infections and infestations) | 7 (7) | 1 (1)
Nasopharyngitis (Infections and infestations) | 13 (15) | 6 (6)
Otitis media (Infections and infestations) | 26 (28) | 9 (10)
Upper respiratory tract infection (Infections and infestations) | 24 (31) | 9 (9)
Cough (Respiratory, thoracic and mediastinal disorders) | 22 (25) | 15 (17)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 5 (5)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 21 (25) | 6 (7)
Rash (Skin and subcutaneous tissue disorders) | 3 (3) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor must have the opportunity to review at least 60 days prior to submission for publication or presentation. If review indicates that potentially patentable subject matter would be disclosed, publication or public disclosure may be delayed for a maximum of an additional 60 days to allow for filing the necessary patent applications